CLINICAL TRIAL: NCT04680559
Title: Influence of a Mindfulness and Compassion-Based Intervention in Psychotherapists: Analysis of Its Effects on Empathy, the Therapeutic Alliance and the Symptomatic Evolution of Their Patients
Brief Title: Mindfulness Training for Psychotherapeutic Care
Acronym: EMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Ausias Cebolla, Full professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 168021
Record Dates: First submitted 2020-11-30; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Mindfulness, Compassion; Empathy, Working Alliance, Patients' Symptomatology, Psychotherapeutic Process; Psychotherapist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCBI Group (Experimental): Training in mindfulness and compassion (MCBI) is facilitated in eight weekly sessions of 2 hours. With a didactic format, through theory, class discussions, and guided meditation practices.
  Interventions: Behavioral: MCBI
- Active-Wait List Group (Active Comparator): Completion of a record during these 8 weeks. Active work of introspection about one's own sensations, thoughts, distractions, judgments, etc. in therapy sessions. Registered after each session.
  Interventions: Behavioral: Active Comparator

INTERVENTIONS:
Behavioral: MCBI — The topics covered in the sessions are: Week 1: Introduction to mindfulness and attention to breathing. Week 2. Open awareness of bodily sensations. Week 3: Work with thoughts, introductory theory and practice in attention to sounds. Week 4: Working with thoughts, advanced theory and practice in mental landscape. Week 5: Introductory theory and practice in labeling emotions. Session 6: Advanced theory in working with emotions and practice in difficult emotions. Week 7: Introductory theory on self-compassion and compassion. Practice in self-compassion. Week 8: Practice in compassion and active compassion (acts of kindness and shared humanity).
  Arms: MCBI Group
Behavioral: Active Comparator — Free observation of the psychotherapist's own feelings, thoughts, distractions, biases and behavior in general for 8 weeks. Observations of these variables are recorded during psychotherapy sessions with patients participating in the research.
  Arms: Active-Wait List Group

SUMMARY:
It has been shown that mindfulness-based interventions (MBI) applied to psychotherapists improve their empathy and increase the therapeutic alliance. It is expected that these improvements may beneficially affect the results of psychotherapy. However, new studies are needed to examine whether an MBI can have an effect on the healthy evolution of these professionals' patients.

The objective of this project is to analyze the influence of a mindfulness and compassion based intervention (MCBI) applied to psychotherapists, on the empathy perceived by their patients, the therapeutic alliance and their symptomatology.

This study is a randomized clinical trial of an intervention based on MBSR and adapted to the population of psychotherapists, including in the last two sessions the practice of compassion, called Mindfulness and Compassion Based Intervention (MCBI). The subjects (n = 63) were randomly assigned to MCBI (n = 33) or to a Waiting List group in which they fill in a self-record of their own feelings, thoughts, etc. in therapy for 8 weeks (n = 30). Participants in the MCBI intervention condition were asked to meet weekly during a two-hour session for two months. Pre / post-intervention and five-month evaluations were performed as a follow-up.

Mindfulness measures (FFMQ) will be taken for the evaluation of psychotherapists, Self-compassion (SCS-SF), negative symptomatology (DASS-21), empathy (EUS-T, TECA), personal therapist style (EPT-C) and mindfulness instructional style (MIQ).

For the evaluation of patients, measures of mindfulness (FFMQ), self-compassion (SCS-SF) will be taken - to try to control without these skills they can be vicariously modified without being directly trained-, subjective well-being (PHI), psychological well-being (BSI), therapeutic alliance (WATOCI, ENAT) and perceived empathy (EUS-P).

DETAILED DESCRIPTION:
The practice of psychotherapy involves the formation and development of a series of skills by the professional. These skills encourage the establishment of a quality therapeutic link, which helps to improve the effectiveness of therapy sessions. In this sense, current research indicates that the link established between the psychotherapist and his patients has a high effect on the evolution and results of psychotherapy. This improvement is to a greater extent attributed to the establishment of the link than to the specific techniques that are applied in therapy.

Among the variables that favor the link, the empathy of the psychotherapist has been widely studied, and has proven to be highly related to the benefits of psychological interventions.

Therefore, the development of healthy empathy is one of the most important variables on which the benefits of psychotherapy are based. It facilitates a true understanding of the vital situations of the patients and is essential in establishing the therapeutic link.

The influence of the latter on the results of psychological interventions has meant that empathy training is one of the basic objectives to follow in the training of clinical and health psychologists, increasing research on effective strategies for this, among which mindfulness and compassion based interventions (MCBI) stand out.

In recent years, the MCBI have established themselves as a very useful intervention in the healthcare field, and several authors suggest the advantages of their application in psychotherapists, pointing out their beneficial influence on the therapeutic relationship and the psychotherapeutic process.

The MCBI are structured interventions in which a series of attitudes and mental states associated with mindfulness and compassion are trained through different meditation techniques. You also learn to generalize these states in the way we relate to the experiences we live. Based on this, the MCBI can be an especially useful strategy to train a series of skills that beneficially influence the therapeutic link and the results of psychotherapy. In relation to the above, it has been seen that MCBI have a beneficial effect on the levels of self-reported empathy of clinical and health psychologists. In addition, an interesting association has been observed between the levels of mindfulness and self-reported empathy in psychotherapists, and between these variables and the therapeutic alliance established with their patients. An association has also been found between the results of the therapeutic alliance measures between therapists and patients after a Mindfulness-based Intervention (MBI). Finally, it has been seen that the application of an MCBI in psychotherapists indirectly influences the evolution of their patients, helping to reduce their symptoms and increase their levels of well-being.

These results imply important support for the advantages of including the MCBI in the training of clinical and health psychologists, in order to increase their levels of empathy and the effectiveness of their interventions. However, there are many limitations we find in these results.

First, the studies that have analyzed the influence of MCBI on empathy only include a self-reported evaluation of psychotherapists on this variable. In addition, this evaluation does not give us information about whether the MCBI affects the empathy that patients perceive in their therapists, which prevents us from assessing whether these benefits exert a real influence on the therapeutic relationship and the psychotherapeutic process.

On the other hand, studies that have established a relationship between levels of mindfulness and direct results in therapeutic alliance include only mindfulness-based interventions (MBI), not including compassion training in a manner explicit. We are interested in observing whether a MCBI significantly influences the perception of the therapeutic alliance by patients.

Finally, in Grepmair's study in which the benefits of applying an MCBI in psychotherapists on the evolution of their patients have been observed, the mediating variables that could explain these results were not evaluated. The objective of this project is to identify the mechanisms of action of the MCBI and its effect on the different variables that could be influencing the results of psychotherapy, such as the empathy of the psychotherapist and the therapeutic alliance established with their patients.

ELIGIBILITY:
Inclusion Criteria:

* Therapists inclusion criteria:

  * Have a psychology degree.
  * Be able to read and write using the Spanish language.
  * Be doing therapy with at least one patient.

Eligible participants were contacted through the main psychotherapeutic schools and university centers to invite them to an explanatory meeting of the study.

* Patient inclusion criteria:

  * Be between 18 and 75 years old.
  * Be able to read and write using the Spanish language.

Eligible participants were contacted by their personal psychotherapist, either by a phone call or regular therapy appointment to invite them to participate in the study.

Exclusion Criteria:

* Therapists exclusion criteria:
* Have extensive experience in mindfulness practice
* Use mindfulness in therapy with your patients.
* Do not engage in clinical psychology or psychotherapy
* Patient exclusion criteria:

  * Serious active mental disorders (schizophrenia, bipolar disorder, psychotic disorders) • Disorders due to active substance use (if consumed in the last year)
  * Cognitive impairment
  * Take more than 2 and a half years in therapy with the same therapist

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in Empathic Understanding Scale Therapist's Version (EUS-TV) | 8 weeks, 6 months
  Designed to assess self-perceived empathy by the therapist himself during therapy sessions. It consists of 16 items and respondents are asked to indicate on a scale of 1 (no, I strongly believe that it is not true) to 6 (yes, I strongly believe that it is true). From this questionnaire a total empathy score is obtained. Higher scores indicate improvements in empathy.
  Used to measure empathy in therapists. EUS has proven effective (Andrade-González, 2009; Barrett-Lennard, 1978)
Empathic Understanding Scale Patient's Version (EUS-PV) | 8 weeks, 6 months
  Designed to assess the empathy of therapists perceived by their patients during therapy sessions. It consists of 16 items and respondents are asked to indicate on a scale of 1 (no, I strongly believe that it is not true) to 6 (yes, I strongly believe that it is true). From this questionnaire a total empathy score is obtained. Higher scores indicate improvements in empathy.
  Used to measure empathy in therapists. EUS has proven effective (Andrade-González, 2009; Barrett-Lennard, 1978)
Changes in Cognitive and Affective Empathy Test (TECA) | 8 weeks, 6 months
  Designed to evaluate self-reported empathy by the therapists themselves. It is made up of 33 items and respondents are asked to indicate on a scale of 1 (totally disagree) to 5 (totally agree). Four subscales are obtained from this questionnaire: perspective adoption, which refers to taking the patient's point of view; emotional understanding; empathic stress, referred to the contagion of the patient's negative emotions; and empathic joy, referring to the ability to feel joy for the positive emotions of others. You also get a total empathy score. Used to measure empathy in therapists.
  TECA has proven effective (López-Pérez, Fernández-Pinto & Abad, 2008)
Changes in Working Alliance Theory of Change Inventory (WATOCI): reduced version of the Therapeutic Alliance Inventory (WAI-S) | 8 weeks, 6 months
  Designed to evaluate the therapeutic alliance, measured by the patient. It is divided into the subscales of tasks, link and joint goals in therapy and Theory of therapist change, with a general measure of therapeutic Alliance. Composed of 17 items with a Likert scale from 1 (Never) to 7 (Always).
  Used to measure therapeutic alliance in patients. WATOCI has proven effective (Corbella & Botella, 2004; Duncan & Miller, 1999).
Changes in Alliance Negotiation Scale (ANS) | 8 weeks, 6 months
  Designed to evaluate the flexibility, negotiation and expression of the therapist measured by the patient. Composed of 12 items with a Likert scale from 1 (Never) to 5 (Often).
  Used to measure therapeutic alliance in patients. ANS has proven effective (Díaz-Oropeza & Peña-Leyva, 2016; Doran, Safran, Waizmann, Bolger & Muran, 2012)
Changes in Brief Sympton Inventory (BSI-18) | 8 weeks, 6 months
  Designed to evaluate somatization, depression and anxiety. Composed of 18 items with a Likert scale from 0 (Nothing) to 4 (A lot).
  Used to measure psychological well-being in patients. BSI-18 has proven effective (Derogatis & Melisaratos, 1983; Ruipérez, Ibáñez, Lorente, Moro & Ortet, 2001)

SECONDARY OUTCOMES:
Changes in Five Facet Mindfulness Questionnaire (FFMQ) | 8 weeks, 6 months
  Designed to evaluate mindfulness capabilities, through the sub-scales of observation, description, acting consciously, not judging one's own experience and not reacting to one's own experience. This short version is composed of 20 items, with a scale ranging from 1 (never or very rarely true) to 5 (very often or always true).
  Used to measure mindfulness in therapists and patients. FFMQ has proven effective (Baer, Smith, Hopkins, Krietemeyer & Toney, 2006; Tran et al., 2014)
Changes in the short scale of self-compassion (SCS-SF) | 8 weeks, 6 months
  Designed to assess common humanity, mindfulness, self-judgment, excessive identification, isolation, personal goodness and general self-compassion. Composed of 12 items in its short version classified on a Likert scale from 1 (almost never) to 5 (almost always) with the total score obtained by adding the averages of each subscale.
  Used to measure self-compassion in therapists and patients. SCS-SF has proven effective (García-Campayo et al., 2014; Raes, Pommier, Neff & Van Gucht, 2011)
Changes in the Mindfulness Instruction Questionnaire (MIQ; adapted from the Mindfulness In Parenting Questionnaire MIPQ) | 8 weeks, 6 months
  Designed to evaluate mindfulness styles in the instruction of therapists and their ability to be present in session. (Obtained from: Mindfulness in Parenting Questionnaire). Composed of 28 items, with a Likert scale from 1 (never) to 5 (almost always).
  Used to measure mindfulness instructional style in therapists. MIPQ has proven effective (McCaffrey, Reitman & Black, 2017)
Changes in Personal Style of the Therapist (PST-Q) | 8 weeks, 6 months
  Designed to evaluate the instructional function, the expressive function, the involvement function, the attentional function and the operative function of the therapist. Composed of 36 items with a Likert scale from 1 (Total disagreement) to 7 (Total agreement).
  Used to measure the therapist's personal style in therapists PST-Q has proven effective (Fernández-Álvarez, García, LoBianco & Corbella, 2003)
Changes in Depression Anxiety Stress Scale (DASS-21) | 8 weeks, 6 months
  Designed to assess levels of depression, anxiety and stress. Composed of 21 items with a Likert scale from 0 (It didn't happen to me) to 3 (It happened a lot, or most of the time) with an overall score obtained from the sum of all the items.
  Used to measure negative symptomatology in therapists. DASS-21 has proven effective (Lovibond & Lovibond, 1993).
Changes in the Pemberton Happiness Index (PHI) | 8 weeks, 6 months
  Designed to assess remembered well-being (divided into the subscales of hedonic well-being, eudaimonic well-being, social well-being and a total score) and experienced well-being (divided into the subscales of positive experiences and experiences negative) Composed of a scale of 12 items that score from 0 to 10 the degree of agreement with each item.
  Used to measure subjective well-being in patients. PHI has proven effective (Hervás & Vázquez, 2013).
Changes in Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) | 8 weeks, 6 months
  Designed to measure the psychotherapeutic process, it evaluates the state of the client or patient from a series of dimensions (subjective well-being, problems / symptoms and general functioning). It is a is a self-report questionnaire composed of 34 items. It also has short forms of 18 (forms A and B), 10 and 5 items to use in each session as a form of continuous monitoring of the therapeutic process. The short form with 5 items was used in this study.
  It consists of a Likert-type scale that goes from 0 (never) to 4 (always or almost always).
  Used to measure the therapeutic process in patients. CORE-OM has been shown to be effective (Evans et al., 2000; Feixas et al., 2012).
Changes in State Emotion Regulation Inventory (SERI) | 8 weeks
  Designed to assess distraction, reassessment, self-criticism and acceptance. Composed of 16 items with a Likert scale from 1 (Strongly disagree) to 7 (Strongly agree).
  Used to measure emotional regulation in therapists. SERI has proven effective (Katz, Lustig, Assis & Yovel, 2017).
Changes in the State-Trait Anxiety Inventory (STAI) | 8 weeks
  Designed to assess the subject's state anxiety, understood as the subjective feelings of tension and apprehension and the hyperactivity of the Autonomous Nervous System. Composed of 20 items on a Likert scale from 0 (Nothing) to 3 (Very good).
  Used to measure anxiety in therapists. STAI has proven effective (Spielberger, Gorsuch & Lushene, 1970).
Changes in Positive and Negative Affect Schedule (PANAS) | 8 weeks
  Designed to assess negative affect and positive affect. Composed of 20 items with a Likert scale from 1 (Very little or nothing) to 5 (Extremely).
  Used to measure affections in therapists. PANAS has proven effective (Sandín et al., 1999; Watson, Clark & Tellegen, 1988).

OTHER OUTCOMES:
Qualitative "Mindfulness and Compassion-Based Intervention" post-training measures | 8 weeks
  Has this training had any effect on your work in therapy? Do you think that the regular practice of mindfulness can provide specific qualities for the exercise of psychotherapy? Have you noticed changes in the way you perceive the feelings or attitudes of your patients? Have you noticed changes in the way you perceive your own feelings, attitudes, thoughts? Do you think that training has been able to affect your way of perceiving biases or interpretations both in yourself and in your patients during therapy? Have you practiced mindfulness, formally or informally, just before a difficult patient entered? Do you think it has helped you in more complex situations in therapy? Have you applied mindfulness with any of your patients? Formally, informally, psychoeducation, modeling? If you could, would you change some of this training?
Quantitative record on "Mindfulness and Compassion-Based Intervention" post-training results | 8 weeks
  Questions Yes / No about psychotherapist training
  Order of mindfulness interest
  Likert scale from 0 (Totally disagree) to 5 (Totally agree) of the MCBI improvements
  Likert scale from 0 (Not very valuable) to 5 (Extremely valuable) Indicate how relevant the different sections of the training have been for you
  Likert scale from 0 (Nothing) to 10 (Very much) Indicate to what degree you believe that the intervention based on mindfulness and compassion that has helped you control aspects that you would previously seek to change or improve.
  Indicate to what degree you notice a global improvement as a result of the intervention you have received.
  Indicate to what degree you have improved in your start-up objectives, as a result of the intervention you have received.
  Questions about Practice and Materials
Qualitative measures post-registration Waiting List Group | 8 weeks
  Did you contribute something to fill in the records? Have you noticed changes in the way you perceive your changes, reactions, distractions...? Have you detected something concrete with any of your patients thanks to having to fill in the records? At what time of the day did you fill in the records? Difficulties when taking records During these last 2 months, have you done any kind of work of introspection, self-knowledge, personal therapy, etc.?
  Observations, something to comment:
Registration of attendance at sessions | 8 weeks
  Weekly record taken by the instructor attending each session.
Record the mindfulness practice between sessions | 8 weeks
  Weekly registration outside the sessions recording: Day of the week, Audio / Type of meditation, minutes of practice, Difficulties / Observations.
Introspective record during therapy sessions Wait List Group | 8 weeks
  It is proposed to carry out a diary or introspective self-registration of what you can happen in therapy sessions with their patients (patients who are participating in this study too). That is, make a weekly record of how it felt The therapist at different times of therapy, providing some examples of changes that can be detected:
  * Distractions of the patient's speech to another topic
  * Postural changes or discomforts (we always talk about you, the therapist)
  * Thoughts and emotions that may arise
  * And in general, anything that wakes you up what your patient says or does
  This registration should be done, if possible, at the end of the session with the patient. If not Possible will be filled that same day at another time.
  In no case will personal data of any of the patients be entered. it is requested to indicate who the patient will be A: your e-mail and B: your e-mail (if you have more than 1).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Garrote Caparrós, Student, Principal Investigator — Universitat de València; Miguel Bellosta Batalla, Dr., Study Director — Universitat de València
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Andrade-González, N. (2009). El papel del terapeuta en la alianza terapéutica. Trabajo presentado en la UNED, Guadalajara, España.
- [Background] Barrett-Lennard, G. T. (1978). The Relationship Inventory: Later developments and adaptations. JSAS: Catalog of Selected Documents in Psychology, 8(68), 1-55
- [Background] Brito, G. (2014). Rethinking mindfulness in the therapeutic relationship. Mindfulness, 5(4), 351-359.
- [Background] Bruce N, Shapiro SL, Constantino MJ, Manber R. Psychotherapist mindfulness and the psychotherapy process. Psychotherapy (Chic). 2010 Mar;47(1):83-97. doi: 10.1037/a0018842. PMID 22402003
- [Background] Corbella, S., & Botella, L. (2004). Psychometric properties of the Spanish version of the Working Alliance Theory of Change Inventory (WATOCI). Psicothema, 16(4), 702-705.
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Díaz-Oropeza, I. F., & Peña-Leyva, L. A. (2016). Validation of the Spanish version of the Therapeutic Alliance Negotiation Scale. Estudios de Psicología, 37(2-3), 604-632.
- [Background] Doran JM, Safran JD, Waizmann V, Bolger K, Muran JC. The alliance negotiation scale: psychometric construction and preliminary reliability and validity analysis. Psychother Res. 2012;22(6):710-9. doi: 10.1080/10503307.2012.709326. Epub 2012 Aug 6. PMID 22861685
- [Background] Duncan, B. L., & Miller, S. D. (1999). Working Alliance Theory of Change Inventory (WATOCI). The Institute for the Study of Therapeutic Change (ISTC)
- [Background] Fernández-Álvarez, H., García, F., LoBianco, J., & Corbella, S. (2003). Assessment questionnaire on the personal style of the therapist PST-Q. Clinical Psychology & Psychotherapy, 10(2), 116-125.
- [Background] Garcia-Campayo J, Navarro-Gil M, Andres E, Montero-Marin J, Lopez-Artal L, Demarzo MM. Validation of the Spanish versions of the long (26 items) and short (12 items) forms of the Self-Compassion Scale (SCS). Health Qual Life Outcomes. 2014 Jan 10;12:4. doi: 10.1186/1477-7525-12-4. PMID 24410742
- [Background] Hervas G, Vazquez C. Construction and validation of a measure of integrative well-being in seven languages: the Pemberton Happiness Index. Health Qual Life Outcomes. 2013 Apr 22;11:66. doi: 10.1186/1477-7525-11-66. PMID 23607679
- [Background] Katz BA, Lustig N, Assis Y, Yovel I. Measuring regulation in the here and now: The development and validation of the State Emotion Regulation Inventory (SERI). Psychol Assess. 2017 Oct;29(10):1235-1248. doi: 10.1037/pas0000420. Epub 2016 Dec 12. PMID 27936820
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Evans, C., Mellor-Clark, J., Margison, F., Barkham, M., Audin, K., Connell, J., & McGrath, G. (2000). CORE: Clinical Outcomes in Routine Evaluation. Journal of Mental Health, 9(3), 247-255.
- [Background] Kiken LG, Garland EL, Bluth K, Palsson OS, Gaylord SA. From a state to a trait: Trajectories of state mindfulness in meditation during intervention predict changes in trait mindfulness. Pers Individ Dif. 2015 Jul 1;81:41-46. doi: 10.1016/j.paid.2014.12.044. PMID 25914434
- [Background] Leonard, H. D., Campbell, K., & Gonzalez, V. M. (2018). The relationships among clinician self-report of empathy, mindfulness, and therapeutic alliance. Mindfulness, 9(6), 1837-1844.
- [Background] López-Pérez, B., Fernández-Pinto, I., & Abad, F. J. (2008). TECA. Test de Empatía Cognitiva y Afectiva. Madrid: Tea Ediciones, S.A.
- [Background] Lovibond, S. H. & Lovibond, P. F. (1993). Manual for the Depression Anxiety Stress Scales (DASS). Psychology Foundation Monograph (Available from The Psychology Foundation, Room 1005 Mathews Building, University of New South Wales, NSW 2052, Australia).
- [Background] McCaffrey, S., Reitman, D., & Black, R. (2017). Mindfulness in Parenting Questionnaire (MIPQ): Development and validation of a measure of mindful parenting. Mindfulness, 8(1), 232-246.
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Ruipérez, M. Á., Ibáñez, M. I., Lorente, E., Moro, M., & Ortet, G. (2001). Psychometric properties of the Spanish version of the BSI: Contributions to the relationship between personality and psychopathology. European Journal of Psychological Assessment, 17(3), 241-250.
- [Background] Ryan A, Safran JD, Doran JM, Muran JC. Therapist mindfulness, alliance and treatment outcome. Psychother Res. 2012;22(3):289-97. doi: 10.1080/10503307.2011.650653. Epub 2012 Mar 15. PMID 22417065
- [Background] Spielberger, C.D., Gorsuch, R.L. and Lushene, R.E. (1970) STAI Manual for the State-Trait Anxiety Inventory. Consulting Psychologists Press, Palo Alto.
- [Background] Tran US, Cebolla A, Gluck TM, Soler J, Garcia-Campayo J, von Moy T. The serenity of the meditating mind: a cross-cultural psychometric study on a two-factor higher order structure of mindfulness, its effects, and mechanisms related to mental health among experienced meditators. PLoS One. 2014 Oct 16;9(10):e110192. doi: 10.1371/journal.pone.0110192. eCollection 2014. PMID 25330072
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Bibeau, M., Dionne, F., & Leblanc, J. (2016). Can compassion meditation contribute to the development of psychotherapists' empathy? A review. Mindfulness, 7(1), 255-263.
- [Result] Grepmair L, Mitterlehner F, Loew T, Bachler E, Rother W, Nickel M. Promoting mindfulness in psychotherapists in training influences the treatment results of their patients: a randomized, double-blind, controlled study. Psychother Psychosom. 2007;76(6):332-8. doi: 10.1159/000107560. PMID 17917468
- [Result] Davis DM, Hayes JA. What are the benefits of mindfulness? A practice review of psychotherapy-related research. Psychotherapy (Chic). 2011 Jun;48(2):198-208. doi: 10.1037/a0022062. PMID 21639664
- [Result] Elliott R, Bohart AC, Watson JC, Murphy D. Therapist empathy and client outcome: An updated meta-analysis. Psychotherapy (Chic). 2018 Dec;55(4):399-410. doi: 10.1037/pst0000175. PMID 30335453
- [Result] Lamothe M, Rondeau E, Malboeuf-Hurtubise C, Duval M, Sultan S. Outcomes of MBSR or MBSR-based interventions in health care providers: A systematic review with a focus on empathy and emotional competencies. Complement Ther Med. 2016 Feb;24:19-28. doi: 10.1016/j.ctim.2015.11.001. Epub 2015 Nov 27. PMID 26860797
- [Result] Nienhuis JB, Owen J, Valentine JC, Winkeljohn Black S, Halford TC, Parazak SE, Budge S, Hilsenroth M. Therapeutic alliance, empathy, and genuineness in individual adult psychotherapy: A meta-analytic review. Psychother Res. 2018 Jul;28(4):593-605. doi: 10.1080/10503307.2016.1204023. Epub 2016 Jul 7. PMID 27389666
- [Result] Norcross, J. C., & Lambert, M. J. (Eds.). (2019). Psychotherapy relationships that work: Volume 1: Evidence-based therapist contributions. New York, NY: Oxford University Press.
- [Result] Schomaker, S. A. (2014). The impact of mindfulness training on therapeutic alliance, empathy, and lived experience: A mixed methods study with counselor trainees. (Dissertation). Texas A&M: University-Corpus